CLINICAL TRIAL: NCT06590272
Title: Comparison on Visual and Refractive Outcomes of Four Different Types of IOL in Patients With Cataracts
Brief Title: Comparison on Outcomes of Four IOLs in Patients With Cataracts
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Sun Yilin, Resident Physician, Shanghai 10th People's Hospital
Other Study IDs: SHSY-LYZX-210
Record Dates: First submitted 2024-08-31; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cataract; Intraocular Lens; Visual Outcomes
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- TECNIS PCB00 IOL (A): The patients in this groups underwent cataract surgery with TECNIS PCB00 IOL
  Interventions: Device: TECNIS PCB00 intraocular lens
- HumanOptics Diff-Aay IOL (B): The patients in this groups underwent cataract surgery with HumanOptics Diff-Aay IOL
  Interventions: Device: HumanOptics Diff-Aay intraocular lens
- TECNIS Symfony ZXR00 IOL (C): The patients in this groups underwent cataract surgery with TECNIS Symfony ZXR00 IOL
  Interventions: Device: TECNIS Symfony ZXR00 intraocular len
- ZEISS AT LISA tri 839MP IOL (D): The patients in this groups underwent cataract surgery with ZEISS AT LISA tri 839MP IOL
  Interventions: Device: ZEISS AT LISA tri 839MP intraocular len

INTERVENTIONS:
Device: TECNIS PCB00 intraocular lens — In this study, we select TECNIS PCB00 IOL for inserting in the eyes during the cataract surgery
  Other Names: IOL
  Groups: TECNIS PCB00 IOL (A)
Device: HumanOptics Diff-Aay intraocular lens — In this study, we select HumanOptics Diff-Aay IOL for inserting in the eyes during the cataract surgery
  Other Names: IOL
  Groups: HumanOptics Diff-Aay IOL (B)
Device: TECNIS Symfony ZXR00 intraocular len — In this study, we select TECNIS Symfony ZXR00 IOL for inserting in the eyes during the cataract surgery
  Other Names: IOL
  Groups: TECNIS Symfony ZXR00 IOL (C)
Device: ZEISS AT LISA tri 839MP intraocular len — In this study, we select ZEISS AT LISA tri 839MP IOL for inserting in the eyes during the cataract surgery
  Other Names: IOL
  Groups: ZEISS AT LISA tri 839MP IOL (D)

SUMMARY:
The objective of this study was to compare the objective visual outcomes and subjective fuctional vision of four different intraocular lens (IOL) in patients underwent cataracts surgery. This was a retrospective study. Patients with age-related cataract underwent phacoemulsification combined with IOLs implantation. Patients were divided into 4 groups. Uncorrected distant visual acuity(UDVA), uncorrected intermediate visual acuity (UIVA), uncorrected near visual acuity (UNVA),and the best corrected visual acuity (BCVA) 1 month and 3 months after the surgery were determined. The defocus curve, contrast sensitivity, and customized VF-14-oriented Visual Function Index questionnaire were performed 3 months postoperatively. Kruskal-Wallis test and generalized estimating equation(GEE) were used to analyze and compare the difference between objective visual outcomes and subjective visual quality among different groups.

DETAILED DESCRIPTION:
The objective of this study was to compare the objective visual outcomes and subjective fuctional vision of four different intraocular lens (IOL) in patients underwent cataracts surgery. This was a retrospective study. Patients with age-related cataract underwent phacoemulsification combined with IOLs implantation. Patients were divided into group A (TECNIS PCB00 IOL), Group B (HumanOptics Diff-Aay IOL), Group C (TECNIS Symfony ZXR00 IOL) and group D (ZEISS AT LISA tri 839MP IOL). Uncorrected distant visual acuity(UDVA), uncorrected intermediate visual acuity (UIVA), uncorrected near visual acuity (UNVA),and the best corrected visual acuity (BCVA) 1 month and 3 months after the surgery were determined. The defocus curve, contrast sensitivity, and customized VF-14-oriented Visual Function Index questionnaire were performed 3 months postoperatively. Kruskal-Wallis test and generalized estimating equation(GEE) were used to analyze and compare the difference between objective visual outcomes and subjective visual quality among different groups.

ELIGIBILITY:
Inclusion Criteria:

* age-related cataract with myopia≤-6.0D and over 0.0D
* axial length≤26mm and corneal astigmatism≤1.5D
* well-cooperation of finishing preoperative examinations
* completion of all follow-up visits

Exclusion Criteria:

* previous eye diseases that affect vision including keratopathy, glaucoma, uveitis, amblyopia, fundus diseases, etc.
* patients with decreased cognitive ability, unable to cooperate with preoperative examination, or suffering from severe anxiety, depression and mental illness
* serious complications during operation, including corneal injury, iris injury, expelling choroidal hemorrhage, posterior capsule rupture, etc
* serious postoperative complications, including displacement of intraocular lens, macular edema, endophthalmitis, etc
* follow-ups less than 3months

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cataract ultrasonic emulsification aspiration with one-stage implantation of 4 types of IOLs at the Shanghai Tenth People's Hospital from October 2021 to June 2023
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative visual acuity | 3 months
  The uncorrected distant visual acuity(UDVA), the best corrected distant visual acuity (BCVA) (5 m), the uncorrected intermediate visual acuity(UIVA) (80 cm) and the uncorrected near visual acuity(UIVA) (40 cm) were chosen as the index to evaluate the VA. The UDVA and BCVA were examined by logarithmic visual acuity chart. The UIVA and UIVA were examined by using a near eye chart.They were all measured 1 month and 3 months after the surgery.
Postoperative contrast sensitivity | 3 months
  The contrast sensitivity was used to conduct the assessment by CSV-1000E (VectorVision, USA) under photopic (85 cd/m2) condition at a 2.5m distance. The logarithmic values for 3, 6, 12, and 18 cycles/degree (c/d) were analyzed 3 months postoperatively.
Postoperative defocus curve | 3 months
  Defocus curve was used to evaluate the visual quality of functional intraocular lens after surgery. The insertion range was -4.0 D ~ + 2.0 D, increasing by 0.5 D. The best corrected distant visual acuity was recorded at each diopter 3 months postoperatively.
Postoperative eye-related quality of life | 3 months after surgery
  Based on the American Questionnaire on Visual Function Index-14 (VF-14), the Chinese-oriented version(VF-12-CN) was used to investigate the postoperative near-vision, visual satisfaction, ocular discomfort, visual disturbance, and subjective feelings of far-vision, middle-vision and near-vision. Each question was divided into 4 levels and the scores ranked from 0 to 3 points. Considering the visual interference such as glare and halo, the evaluation of glare and halo visual interference phenomenon was also added.

CONTACTS AND LOCATIONS:
Overall Officials: Yiwen Hu, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China